CLINICAL TRIAL: NCT03152968
Title: Proficiency of Fundamental Movement Skills in 5 -10 Years Old School Children in Udupi District
Brief Title: To Observe Ability of Fundamental Movement Skills in School Children of Age 5 to 10-year-old in Udupi District
Acronym: FMS
Status: Completed | Type: Observational
Sponsor: Manipal University (Other)
Responsible Party: Principal Investigator, Mayuri Gad, Postgraduate student, Manipal University
Other Study IDs: REF/2017/05/014215
Record Dates: First submitted 2017-05-09; First posted 2017-05-15 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Physical Activity
Keywords: FMS
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fundamental movement skill is the precursor for physical activity in later life. Proficiency of Fundamental Movement Skills in Indian School Children is unknown. This observational trial shall tell us how proficient are our Udupi District Children.

DETAILED DESCRIPTION:
After IRC and IEC approval and approval from district educational officers, proper assent and consent will be given to the principal of the respective school.

1-week prior to the study, parents will be explained about the study during parent meeting and even school leaving and opening times, a parent who visits the school to drop their children will be addressed.

Children of age above 7 yr. will be explained the class about the study.

Inform sheets will be distributed after conveying the information.

Only the children who get an informed sheet signed will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* All children in the age group 5 to 10 year old

Exclusion Criteria:

* Cerebral palsy
* Attention deficit/hyperactivity disorder
* Autism

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children between age 5 to 10 years going to school in Udupi district, who will get consent sign from the parent will be included.
Sampling Method: Probability Sample
Enrollment: 461 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Fundamental movement skill score | immediate
  Satisfying the criterion of each skill such as run, jump, catch, throw

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Sport Science Medicine and Research, Udupi, Karnataka, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mukherjee S, Ting Jamie LC, Fong LH. Fundamental Motor Skill Proficiency of 6- to 9-Year-Old Singaporean Children. Percept Mot Skills. 2017 Jun;124(3):584-600. doi: 10.1177/0031512517703005. Epub 2017 Apr 4. PMID 28376671
- [Result] Birch S, Cummings L, Oxford SW, Duncan MJ. Examining Relative Age Effects in Fundamental Skill Proficiency in British Children Aged 6-11 Years. J Strength Cond Res. 2016 Oct;30(10):2809-15. doi: 10.1519/JSC.0000000000000526. PMID 24832979
- [Result] Morgan PJ, Barnett LM, Cliff DP, Okely AD, Scott HA, Cohen KE, Lubans DR. Fundamental movement skill interventions in youth: a systematic review and meta-analysis. Pediatrics. 2013 Nov;132(5):e1361-83. doi: 10.1542/peds.2013-1167. Epub 2013 Oct 28. PMID 24167179